CLINICAL TRIAL: NCT04267341
Title: Examining The Change of Upper and Lower Extremity Skills With The Effect of Dual Task in Parkinson's Disease Patients
Brief Title: Effect of Dual Task on Upper and Lower Extremity Skills in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elvan ÖZCAN GÜLŞEN, Principal Investigator, Hacettepe University
Other Study IDs: 2019/24-01
Record Dates: First submitted 2020-02-11; First posted 2020-02-12 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Stage Parkinson's Disease Patients: Modified Hoehn and Yahr stage 1-2
  Interventions: Other: Timed Up and Go Test; Other: 10 Meter Walk Test; Other: Purdue Pegboard Test
- Moderate Stage Parkinson's Disease Patients: Modified Hoehn and Yahr stage 2.5-3
  Interventions: Other: Timed Up and Go Test; Other: 10 Meter Walk Test; Other: Purdue Pegboard Test
- Healthy Control: Healthy People
  Interventions: Other: Timed Up and Go Test; Other: 10 Meter Walk Test; Other: Purdue Pegboard Test

INTERVENTIONS:
Other: Timed Up and Go Test — It requires individual to stand up from an armed chair, walk 3m, turn around, walk back to the armed chair, and sit down again
Other: 10 Meter Walk Test — 10 Meter Walk Test measures the time required to complete straight walk of 10 meters distance
Other: Purdue Pegboard Test — Purdue Pegboard test evaluates the fine manuel dexterity

SUMMARY:
The aim of the study is to investigate the change of lower and upper extremity skills with dual task in Parkinson's disease patients and to determine the differences between Parkinson's disease patients with different stages of disease and the healthy controls regarding the change of lower and upper extremity skills with dual task.

ELIGIBILITY:
Inclusion Criteria:

* Modified Hoehn & Yahr (H&Y) stages 1 to 3
* at least 40 years of age
* 21 or more MoCA score.

Exclusion Criteria:

* other neurologic disorder
* any orthopedic problem that could prevent to participate in the study
* severe dyskinesia or tremor
* visual or speech problems

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who apply to the Hacettepe University, Faculty of Physiotherapy and Rehabilitation, Department of Neurological Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | 10-15 seconds
  Functional mobility is assessed by using the timed up and go test. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.
10 Meter Walk Test | 10-15 seconds
  10 Meter Walk Test measures the time required to complete straight walk of 10 meters distance.
Purdue Pegboard Test | 3-5 minutes
  Purdue Pegboard Test assesses the speed and motor dexterity of each hand and the manual dexterity using both hands at the same time. The PPT consists of a board with two columns with 25 holes each and a specific number of pins, washers and collars placed in four containers across the top of the board.

SECONDARY OUTCOMES:
Modified Hoehn and Yahr Scale | 1 minute
  Modified Hoehn and Yahr Scale allocates stages from 0 to 5 to indicate the relative level of disability and stage of disease. Higher level indicates worse physical condition.
Montreal Cognitive Assessment (MoCA) | 10-15 minutes
  Montreal Cognitive Assessment (MoCA) will be used in order to evaluate cognition. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.It' score ranged from 0 to 30 and higher points indicates better cognitive outcomes.
Short-Form 8-Item Parkinson's Disease Questionnaire (PDQ-8) | 1-2 minutes
  The short-form 8-item Parkinson's disease Questionnaire (PDQ-8) is the most commonly used scale measuring health related quality of life (HRQoL) in PD patients. It includes 8 items, and each item has five options (never, occasionally, sometimes, often, always or cannot do at all). The total score ranges from 0 to 32. Higher scores indicates poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No